CLINICAL TRIAL: NCT03237793
Title: Treatment of Hypersensitivity Using Diode Laser and Potassium Nitrate Desensitising Agent- a Comparison of Treatment Effects on Fluorosed and Non-fluorosed Teeth- an in Vivo Randomised Controlled Trial
Brief Title: Treatment of Hypersensitivity Using Diode Laser and Desensitising Agent on Fluorosed and Non-fluorosed Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_45912
Record Dates: First submitted 2017-07-26; First posted 2017-08-03 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Fluorosis, Dental; Non-Fluoride Enamel Opacities; Dentin Sensitivity
MeSH Terms: conditions — Fluorosis, Dental; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: The present study was designed as a randomised controlled clinical trial which was unicenter, double-blinded, parallel designed study, according to the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.
Who Masked: Participant, Outcomes Assessor
Masking Description: A unified stratified randomization, double blind controlled parallel designed was the type generated the allocation sequence. A skilled assistant enrolled the participants and assigned the participants to interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorosed Group (Active Comparator): 45 patients for the fluorosis groupGROUP 1A: Patients with healthy fluorosed teeth receiving desensitising agent (potassium nitrate- RA Themoseal**) treatment. (n=15) GROUP 1B: Patients with healthy fluorosed teeth receiving diode laser treatment$. (n=15) GROUP 1C: Patients with healthy fluorosed teeth receiving diode laser + desensitising agent (potassium nitrate- RA Thermoseal**) treatment. (n=15)
  Interventions: Procedure: Fluorosed Group
- Non Flourosed Group (Placebo Comparator): 45 patients for the non-fluorosis groupGROUP 2- Non Flourosed Group (n=45) GROUP 2A: Patients with healthy non fluorosed teeth receiving desensitising agent (potassium nitrate- RA Thermoseal**) treatment. (n=15) GROUP 2B: Patients with healthy non fluorosed teeth receiving diode laser treatment. (n=15)GROUP 2C: Patients with healthy non fluorosed teeth receiving diode laser + desensitising agent (potassium nitrate- RA thermoseal**) treatment. (n=15
  Interventions: Procedure: Non Flourosed Group

INTERVENTIONS:
Procedure: Fluorosed Group — A single episode of laser therapy with without potassium nitrate (RA Thermoseal*) desensitising agent application was administered to the patients, A group only with desensitising paste and A group with desensitising paste and laser treatment depending on the study group they were assigned
  Arms: Fluorosed Group
Procedure: Non Flourosed Group — A single episode of laser† therapy with or without potassium nitrate (RA Thermoseal*) desensitising agent application was administered to the patients, depending on the study group they were assignedGROUP 2B: Patients with healthy non fluorosed teeth receiving diode laser treatment$. (n=15)GROUP 2C: Patients with healthy non fluorosed teeth receiving diode laser + desensitising agent (potassium nitrate- RA thermoseal**) treatment.
  Arms: Non Flourosed Group

SUMMARY:
The present study was designed as a randomised controlled clinical trial which was unicenter, double-blinded, parallel designed study, according to the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010. The study period was from July 2014 to September 2015.

DETAILED DESCRIPTION:
90 Patients visiting the Out Patient of Department of Periodontology, Krishnadevaraya College of Dental Sciences and Hospital, Bengaluru, India, presenting with a chief complaint of dentinal hypersensitivity were enrolled in the study. Patients' age ranged from 18-60 years. The subjects interested in participating were explained in detail the treatment protocol. A verbal consent as well as a written informed consent was obtained from each patient Treatment of dentinal hypersensitivity with a combination of diode laser and potassium nitrate desensitising agent was considered as the test group and this was compared with diode lasers alone and desensitising agent alone as the positive control groups. The study was conducted in full accordance with the declared ethical principles (World Medical Association Declaration of Helsinki, version VII, 2013)13 and was approved by the Institutional review board of Krishnadevaraya College of Dental Science and Hospital, under the registration number of (ACA/DCD/SYN/KCODS - B/PG/2013-2014).

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a positive response for hypersensitivity testing (Pashley, 1990) i.e. cold water testing using ice cold water (Trowbridge et al., 1980),

  * Air blow test (Coleman and Kinderknecht, 2000),
  * Electric tactile stimulation test (Camps and Pashley, 2003),
  * Patients presenting with non-carious cervical lesions in the enamel (Loomba et al., 2013), fluorosed teeth wherein fluorotic enamel staining confirmed by clinical examination, healthy non fluorosed teeth, which was confirmed by clinical examination (Dean, 1934).

Exclusion Criteria:

* The following were set as the exclusion criteria;

  * Patients undergoing any form of restorative endodontic,
  * Orthodontic treatment or crown restorations,
  * Local defects including caries and fractures,
  * Presence of any systemic diseases,
  * Acute pain conditions (like apical periodontitis, periapical abscess),
  * Presence of periodontal disease or a history of periodontal treatment in last 6 months,
  * Usage of desensitising toothpaste or mouth rinse in the last 4 weeks,
  * Patients allergic to ingredients used in the study product,
  * Teeth with intrinsic stains caused by other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reduction in hypersensitivity | 30 minutes
  The primary outcome that was assessed in the study was the reduction in dentinal hypersensitivity sensation. The visual analogue scale was used as a recording scale when tested with the tests for hypersensitivity, which were the testing with a blast of air, ice cold water testing and electrical tactile sensitivity testing using a scratch-o-meter.

SECONDARY OUTCOMES:
use of diode laser in reducing hypersensitivity | 30 mins
  Efficacy of treatment when diode laser is used alone as a treatment option after scaling and root planing.
use of desensitising agent alone | 30 minutes
  Efficacy of treatment when desensitising agent was used as monotherapy after scaling and root planing
combination of densensitising agent and diode laser | 30 minutes
  3. Efficacy of treatment when a combination of diode laser and desensitising agent was used after scaling and root planing, for the treatment of dentinal hypersensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Paramashivaiah, MDS, Principal Investigator — Krishnadevaraya college of dental sciences